CLINICAL TRIAL: NCT03440255
Title: Transcutaneous Vagus Nerve Stimulation (TaVNS) in Private Healthcare Center: An Open-Label, Non-Randomized Feasibility Study Targeting Anxiety, Chronic Pain and Irritable Bowel Syndrome
Brief Title: Transcutaneous Vagus Nerve Stimulation in Private Healthcare Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kinesis Health Associates (Other)
Responsible Party: Principal Investigator, Pascal J.D. Grolaux, DO, Principal Investigator, Kinesis Health Associates
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TaVNS_PHC
Record Dates: First submitted 2018-02-01; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Generalized Anxiety Disorder; Chronic Pain; Irritable Bowel Syndrome
Keywords: Transcutaneous Vagus nerve Stimulation; Generalized Anxiety Disorder; Chronic Pain; Irritable Bowel Syndrome; Private Practice
MeSH Terms: conditions — Generalized Anxiety Disorder; Chronic Pain; Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transcutaneous Vagus Nerve Stimulation (Experimental): TaVNS 8 sessions, 30 min, 4 weeks GAD: 20 Hertz (Hz) - 80 microseconds (µs) CP: 5Hz-200µs IBS: 3Hz-250µs
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Vagus Nerve Stimulation — TaVNS will be applied by the TENS 7000 device. The stimulation was set according the group of treatment: (GAD: 20Hz-80µs), (CP: 5Hz-200 µs), (IBS: 3Hz-250µs).
  The current intensity was individually established under the pain threshold .The stimulus generates an continous asymmetric biphasic waveform. Ear clip electrodes were plugged in the concha area of the left ear. The stimulation will last 30 min per session (total=8)

SUMMARY:
This non-randomized, open-label study has the objective to study the effects and feasibility of Transauricular Vagus Nerve Stimulation (TaVNS) for patients suffering from Generalized Anxiety Disorder (GAD), Chronic Pain (CP) and Irritable Bowel Syndrome (IBS) in a private healthcare centre.

DETAILED DESCRIPTION:
The effects of TaVNS on GAD, CP and IBS. Participants were investigated during a 4-week period and a 2-month follow-up. Groups (GAD, CP, IBS) were assessed using questionnaires: Anxiety (Generalized Anxiety Disorder GAD-7); CP (Brief Pain Inventory Short Form Questionnaire) and IBS (Irritable Bowel Syndrome Severity Scoring System). TaVNS was performed using a standard transcutaneous electrical nerve stimulation (TENS) device and ear clip electrodes plugged into the concha area of the left ear. All participants received a bi-weekly 30 minutes stimulation (8 sessions). We defined three different TaVNS parameters for each group in hertz (Hz) and microsecond (µs), (GAD: 20Hz-80µs), (CP: 5Hz-200 µs), (IBS: 3Hz-250µs).

ELIGIBILITY:
Inclusion Criteria:

1. Age range 20-65 years old
2. Patient suffering from either Generalized Anxiety Disorder, Chronic Pain scoring and Irritable Bowel Syndrome from moderate
3. Patients meet the scoring standard questionnaires: mild to severe
4. Patient can understand and answer the questions
5. Patient exhibits symptoms for at least six months

Exclusion Criteria:

1. Reading difficulties
2. Diagnosed left ear lesion
3. Measured blood pressure under 100/60 with or without anti-high blood pressure medicine
4. Active implant such as cochlear implant
5. Wounds and skin disease in the left ear
6. Recent head trauma or concussion
7. Cardiac pacemaker
8. Severe alcoholism
9. Left cervical vagotomy
10. Cholinergic or B blocking medicine
11. Recreative drugs
12. Diagnosed concomitant psychiatric comorbidity
13. Diagnosed concomitant personal disorders
14. Diagnosed pregnancy
15. Diagnosed concomitant severe neurological or medical diseases such as neoplasms in activity, neurodegenerative diseases and chronic infectious diseases uncompensated

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline generalized anxiety disorder severity | baseline, 4-week and 2-month follow-up
  To assess the response effect of the TaVNS on the severity of anxiety disorders measured by the 21 items self-administered Generalized Anxiety Disorder GAD-7 questionnaire, where scoring scores of 5, 10 and 15 represent cut-off points for mild, moderate and severe anxiety. A response will be considered as a reduced cut-off point from baseline.
Change from baseline pain severity and pain interference | baseline, 4-week and 2-month follow-up
  To assess the response effect of the TaVNS on the severity of pain and the impact of this pain on daily functioning (Interference) measured by the 9 items self-administered Brief Pain Inventory (Short Form) questionnaire; from 0 (no pain) to 10 (worst pain), ratings from 1 to 4 corresponded to mild pain, 5 to 6 to moderate pain, and 7 to 10 to severe pain with cut-off points being 4 and 6. Scoring pain severity is the mean of the total pain score out of 10. Interference from 0 (no interference) to 10 (completely interferes), rating mild (<=5), moderate (6-7), and severe (>= 8) with cut-off points being 5 and 7. Scoring the interference severity is the mean of the total Interference score out of 10. A response will be considered as a reduced cut-off point from baseline.
Change from baseline irritable bowels syndrome severity | baseline, 4-week and 2-month follow-up
  To assess the response effect of the TaVNS on the severity of irritable bowel syndrome measured by the self-administered Irritable Bowel Syndrome Severity Scoring System (IBS-SSS), where the maximum achievable score is 500. Mild, moderate and severe categories were indicated by scores of 75 to 175, 175 to 300 and > 300 respectively, with cut-off points being 175 and 300. A response will be considered as a reduced cut-off point from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal JD Grolaux, DO, Principal Investigator
Locations (1):
- Kinesis Health Associates, Dartmouth, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salim S, Chugh G, Asghar M. Inflammation in anxiety. Adv Protein Chem Struct Biol. 2012;88:1-25. doi: 10.1016/B978-0-12-398314-5.00001-5. PMID 22814704
- [Background] Bonaz B, Picq C, Sinniger V, Mayol JF, Clarencon D. Vagus nerve stimulation: from epilepsy to the cholinergic anti-inflammatory pathway. Neurogastroenterol Motil. 2013 Mar;25(3):208-21. doi: 10.1111/nmo.12076. Epub 2013 Jan 29. PMID 23360102
- [Background] Nagarajan L, Walsh P, Gregory P, Lee M. VNS therapy in clinical practice in children with refractory epilepsy. Acta Neurol Scand. 2002 Jan;105(1):13-7. doi: 10.1034/j.1600-0404.2002.00129.x. PMID 11903103
- [Background] Trevizol AP, Taiar I, Barros MD, Liquidatto B, Cordeiro Q, Shiozawa P. Transcutaneous vagus nerve stimulation (tVNS) protocol for the treatment of major depressive disorder: A case study assessing the auricular branch of the vagus nerve. Epilepsy Behav. 2015 Dec;53:166-7. doi: 10.1016/j.yebeh.2015.10.002. Epub 2015 Nov 12. No abstract available. PMID 26580212
- [Background] Napadow V, Edwards RR, Cahalan CM, Mensing G, Greenbaum S, Valovska A, Li A, Kim J, Maeda Y, Park K, Wasan AD. Evoked pain analgesia in chronic pelvic pain patients using respiratory-gated auricular vagal afferent nerve stimulation. Pain Med. 2012 Jun;13(6):777-89. doi: 10.1111/j.1526-4637.2012.01385.x. Epub 2012 May 8. PMID 22568773
- [Background] Bonaz B, Sinniger V, Pellissier S. The Vagus Nerve in the Neuro-Immune Axis: Implications in the Pathology of the Gastrointestinal Tract. Front Immunol. 2017 Nov 2;8:1452. doi: 10.3389/fimmu.2017.01452. eCollection 2017. PMID 29163522
- [Result] George MS, Ward HE Jr, Ninan PT, Pollack M, Nahas Z, Anderson B, Kose S, Howland RH, Goodman WK, Ballenger JC. A pilot study of vagus nerve stimulation (VNS) for treatment-resistant anxiety disorders. Brain Stimul. 2008 Apr;1(2):112-21. doi: 10.1016/j.brs.2008.02.001. Epub 2008 Mar 28. PMID 20633378